CLINICAL TRIAL: NCT00588679
Title: Magnetic Resonance Spectroscopic Imaging of the Prostate at 3 Tesla
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-035
Record Dates: First submitted 2007-12-24; First posted 2008-01-08 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Prostate Cancer; MRI
Keywords: Prostate Cancer; Cancer; MRI; Magnetic Resonance Imaging; 06-035
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Magnetic Resonance Spectroscopy

ARMS (1):
- 1 (Experimental): Patients taking part in this study will have one MRI and one MRSI scan acquired in succession during a single MR examination. For those patients who have undergone prostate biopsy it is recommended that this should be done at least eight weeks after the prostate biopsy and should take one hour to one hour and ten minutes total to complete.
  Interventions: Other: Magnetic Resonance Imaging; Spectroscopic Imaging, Contrast Enhanced Imaging

INTERVENTIONS:
Other: Magnetic Resonance Imaging; Spectroscopic Imaging, Contrast Enhanced Imaging — All MR examinations will be performed on a 3.0 Tesla whole body GE MR scanner located at the main campus (1275 York Avenue) or the Breast and Imaging Center (BAIC)(located on Second Ave. between 65th and 66th Streets). The MR examination will include MR imaging and spectroscopic imaging employing a combined torso phased array and endorectal coil receiver. The examination will require one hour to one hour and ten minutes.
  Other Names: MRI

SUMMARY:
The purpose of this study is to determine the benefits of Magnetic Resonance Imaging (MRI) combined with Magnetic Resonance Spectroscopic Imaging (MRSI), on an instrument called a 3.0 Tesla (T) MR scanner.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have clinically suspected or biopsy proven prostate cancer. If a patient has been diagnosed with prostate cancer an official report of biopsy from MSKCC or outside site is required. All outside pathology reports will be confirmed at MSKCC.
* For those patients who have undergone prostate biopsy it is recommended that the interval between biopsy and protocol MRI/MRSI should be at least 8 weeks.
* Patient is a potential surgical candidate for treatment of prostate cancer
* Patient is willing to undergo an endorectal MRI/MRSI exam on the 3.0T MR scanner

Exclusion Criteria:

* Patients who because of general medical or psychiatric condition, or physiologic status unrelated to the presence of prostate cancer cannot give valid informed consent.
* Patients who are unwilling or unable to undergo MRI/MRSI (including patients with contra-indications to MRI such as the presence of cardiac pacemakers or non-compatible intracranial vascular clips.
* Patients who cannot tolerate or have contra-indications to endorectal coil insertion; for example, patients who have had a prior abdominoperineal resection of the rectum or have Crohn's disease, patients with severe hemorrhoids, patients who have had prior radiation to the pelvis to treat a malignancy, or patients who have had minor rectal surgery within the previous 8 weeks.
* Patients with an allergic reaction to latex.
* Patients with a metallic hip implant or any other metallic implant or device in the pelvis that might distort local magnetic field and compromise quality of MRI/MRSI.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2006-08-22 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

PRIMARY OUTCOMES:
To define the relative proton metabolite levels detected by MRSI at 3.0 T in normal and cancerous tissue using pathology as the gold standard. | 3 years

SECONDARY OUTCOMES:
To measure the sensitivity and specificity of localized detection of prostate cancer by 3.0 T MRSI using pathology as the gold standard. | 3 years
To explore whether metabolic markers measured by 3.0 T MRSI are correlated with prostate cancer aggressiveness as defined by the Gleason score. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yousef Mazaheri-Tehrani, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering web site — http://www.mskcc.org